CLINICAL TRIAL: NCT04207073
Title: The Effect of Median Nerve Mobilization on Two Point Discrimination
Brief Title: Assessment of Two Point Discrimination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Gülay Aras, PhD PT, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10840098-604.01.01-E.63690
Record Dates: First submitted 2019-12-14; First posted 2019-12-20 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Assessment, Self
Keywords: two-point discrimination; neural mobilization; tactile sensation; median nerve

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No intervention.
- Exercise group (Experimental): Participants in the exercise group will perform 2 sets of 5 repetitive Median nerve mobilization exercises (total of 20 sessions) per day for 10 days.
  Interventions: Device: Mobilization of median nerve

INTERVENTIONS:
Device: Mobilization of median nerve — Neural mobilization
  Arms: Exercise group

SUMMARY:
When the studies in the literature are examined, no study has been reached to examine whether median nerve mobilization causes changes in two-point discriminatory values in healthy individuals. This study aimed to investigate the effect of median nerve mobilization exercise on two-point discrimination in healthy adult male and female participants. Secondly, it was aimed to determine the role of variables such as gender, age, BMI (weight in kilograms, height in meters and weight and height will be combined to report BMI in kg/m^2), smoking, dominant extremity and physical activity level in 2-point discrimination.

DETAILED DESCRIPTION:
Two-point discrimination is one of the most important cortical senses that require strong tactile sensitivity and the ability to distinguish two points from one point on the skin. Neural mobilization has been reported to be effective in the nerve-related waist, leg, neck, arm, and plantar heel pain, but there is still insufficient evidence for other neuromusculoskeletal problems. It has been stated that factors such as application technique, type and patient characteristics of mobilization are effective in the treatment and more comprehensive studies should be done on this subject. This study aimed to investigate the effect of median nerve mobilization exercise on two-point discrimination in healthy adult male and female participants.

120 healthy female and male adult individuals (60 females, 60 males) will be included in the study. Individuals will be divided into two groups as female and male (n = 60), and a two-point discrimination test will be performed on the palmar face of both hands from the distal phalanx, forefinger, middle finger and palm. After the evaluation, the participants in both groups were randomly divided into two groups as the exercise group (n = 30) and control group (n = 30). Participants in the exercise group will perform 2 sets of 5 repetitive Median nerve mobilization exercises (total of 20 sessions) per day for 10 days. After the exercise program, the two-point discrimination measures will be repeated in all groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers
* Adapt to median nerve mobilization exercise

Exclusion Criteria:

* Upper extremity neuromuscular disease
* The presence of neurological disease
* Skin diseases (burn or scar tissue in upper extremity)
* Diabetes mellitus

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 60 females, and 60 males
Enrollment: 120 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2021-04-24 (Actual); Study Completion 2021-06-26 (Actual)

PRIMARY OUTCOMES:
Two-point discrimination | 2 weeks
  Two-point discrimination test will be performed on the palmar face of both hands from the distal phalanx, forefinger, middle finger and palm.

CONTACTS AND LOCATIONS:
Overall Officials: Candan Algun, Prof., Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No